CLINICAL TRIAL: NCT00061204
Title: Functional Neuroimaging of Social Cognitive and Emotional Processing: Technical and Cognitive Issues
Brief Title: Magnetic Resonance Imaging of the Brain in Emotional Processing
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030195; 03-N-0195
Record Dates: First submitted 2003-05-21; First posted 2003-05-22 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-04

CONDITIONS: Healthy
Keywords: fMRI; Susceptibility Artifacts; Prefrontal Cortex; Temporal Lobes; Methodology; Healthy Volunteer; HV

SUMMARY:
This study will use magnetic resonance imaging (MRI) to identify brain regions involved in performing certain tasks, especially those involving emotions. MRI is a diagnostic tool that uses a strong magnetic field and radio waves to produce images of structural and chemical changes in the brain. The study will also examine which MRI techniques are best to use when scanning brain areas involved in different emotions.

Healthy normal volunteers between 18 and 40 years of age who are right-handed and are native English speakers may be eligible for this study. Individuals with a history of neurological disease, post-traumatic stress disorder or other psychiatric disorder, or who have a history of physical or sexual abuse may not participate. Candidates will be screened with a written questionnaire and a medical history, including psychiatric and neurological information.

Participants will perform tasks involving emotions while undergoing MRI scanning. For this procedure, the subject lies on a table in a narrow metal cylinder (the scanner) containing a magnetic field. Scanning time varies from 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. The subject is asked to lie still for up to 10 minutes at a time. During the scan, the subject performs simple tasks involving the viewing of pictures on a screen. Other tasks involve viewing pictures and responding to them by pressing buttons. Some pictures are violent or pornographic, while others are pleasant to view. Of a total of 162 pictures, 30 percent are categorized as graphic and possibly disturbing.

DETAILED DESCRIPTION:
The purpose of the protocol is to localize the neural regions and systems mediating the forms of knowledge representations hypothesized by the principal investigator to be stored in the human prefrontal cortex. Utilizing experimental neuropsychological tasks during functional MRI on healthy adult volunteers, we will investigate hypotheses regarding the role of the ventromedial prefrontal cortex in social cognition and emotional processing as opposed to the dorsolateral prefrontal cortex, involved in nonsocial-events (planning, problem solving, economic exchange and reasoning). We will also attempt to determine the relationship between non-frontal neural structures involved in emotional expression, such as the amygdala, and those frontal neural structures involved in executive functions that may modulate emotion. Another goal of our study is to test different fMRI sequences to determine which one gives us the best quality of signal in the amygdala and orbitofrontal cortex (affected by signal drop-out due to magnetic susceptibility artifacts). The data that we collect in this protocol will be of value in (1) identifying a set of neural regions and distributed networks mediating the forms of knowledge representation stored in the prefrontal cortex, and (2) contributing to optimization of functional imaging of the amygdala and orbitofrontal cortex at high field strength (3 Tesla). We will also use the data obtained in these studies to constrain theories of frontal lobe function and to provide evidence for the role of specific frontal cortex sectors in specific cognitive functions.

ELIGIBILITY:
INCLUSION CRITERIA:

The study population will consist of young healthy volunteers.

Age range: 18 to 40

Right-handedness (some left-handed subjects may be recruited for preliminary behavioral studies)

EXCLUSION CRITERIA:

Individuals with a neurological or psychiatric history or medical condition that would compromise our interpretation of the fMRI results will be excluded.

Individuals with a current or past history of post-traumatic stress disorder or other psychiatric disorder or individuals with a history of physical or sexual abuse will be excluded as they may be disturbed by viewing graphic pictures.

Subjects with contraindications to exposure to high magnetic field.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38
Dates: Start 2003-05; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Belliveau JW, Kennedy DN Jr, McKinstry RC, Buchbinder BR, Weisskoff RM, Cohen MS, Vevea JM, Brady TJ, Rosen BR. Functional mapping of the human visual cortex by magnetic resonance imaging. Science. 1991 Nov 1;254(5032):716-9. doi: 10.1126/science.1948051.
- [Background] Belliveau JW, Rosen BR, Kantor HL, Rzedzian RR, Kennedy DN, McKinstry RC, Vevea JM, Cohen MS, Pykett IL, Brady TJ. Functional cerebral imaging by susceptibility-contrast NMR. Magn Reson Med. 1990 Jun;14(3):538-46. doi: 10.1002/mrm.1910140311. PMID 2355835
- [Background] Bodner M, Kroger J, Fuster JM. Auditory memory cells in dorsolateral prefrontal cortex. Neuroreport. 1996 Aug 12;7(12):1905-8. doi: 10.1097/00001756-199608120-00006. PMID 8905689